CLINICAL TRIAL: NCT00386646
Title: A Comparative Study of 0.5% Carboxymethylcellulose With 0.005% Stabilized Oxychlorocomplex (PURITE™) Versus 0.5% Carboxymethylcellulose in the Treatment of Dry Eye: A Randomized Controlled Trial
Brief Title: Comparative Study of 0.5% Carboxymethylcellulose With 0.005% Stabilized Oxychlorocomplex (PURITE™) Versus 0.5% Carboxymethylcellulose in the Treatment of Dry Eye
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 152/2004
Record Dates: First submitted 2006-10-10; First posted 2006-10-11 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2006-10

CONDITIONS: Dry Eye Syndromes
Keywords: Dry eye syndromes therapy
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Carboxymethylcellulose Sodium; MCC protocol

INTERVENTIONS:
Drug: 0.5% carboxymethylcellulose (CMC) with purite and CMC alone

SUMMARY:
To compare if 0.5% carboxymethylcellulose with 0.005% SOC (Stabilized oxychloro complex) have the same effectiveness and safety as 0.5% carboxymethylcellulose on dry eye patients.

DETAILED DESCRIPTION:
Dry eye is the very common disorder of tear film. There are millions of people who have dry eye around the world. Dry eye patients may suffer from redness, sandy sensation, itching, excessive watering, burning sensation, excessive mucous discharge, blurred vision, contact lens intolerance, and increased risk of ocular surface damage and ocular infection. Currently, there is no curative treatment for dry eye. The mainstay of treatment is still artificial tear supplement or punctual occlusion. In moderate to severe dry eye patients, the standard replacement is using non-preservative artificial tear more than 4 times a day. However, non-preservative artificial tear has some limitation such as inconvenience to carry, expensive, ocular surface trauma due to sharp plastic tip.

Recently, there is improvement in using new disappearing preservatives in artificial tears. One of the new preservative is stabilized Oxychlorocomplex (SOC, Purite™) which can dissipate into water and sodium chloride, components of natural tears when exposed to light. It also has bactericidal and viricidal activities. Scanning electron microscopy also reveals that, carboxymethylcellulose (CMC) with SOC has a very low toxicity to corneal epithelium than other preservative.

The past study had documented that 0.5% CMC preserved with SOC was safe, comfortable and well tolerated for mild to moderate dry eye patients when applying 4-8 times daily.

The objective of this study was comparing efficacy, tolerability, and safety of 0.5% carboxymethylcellulose(CMC) with Stabilized Oxychlorocomplex(SOC) and 0.5% carboxymethylcellulose alone in patients with moderate to severe dry eye symptoms and/or signs.

ELIGIBILITY:
Inclusion Criteria:

* Out patients of Ophthalmology department, King Chulalongkorn Memorial Hospital, who have symptoms and/or signs of dry eye
* Bilateral dry eye symptoms and/or signs with equal severity between both eyes
* Age > 18 years, capable of following the study protocol, and considered be able to return for all scheduled visit

Exclusion Criteria:

* Different severity of dryness between both eyes
* Current or recent use of topical ophthalmic medications that could affect dry eye condition
* History of any systemic or ocular disorder or condition that could possibly interfere with the interpretation of study result
* Recent contact lens wear (within one month)
* Known hypersensitivity to 0.005% SOC or carboxymethylcellulose
* Pregnancy or planned pregnancy
* Having received permanent punctal occlusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2004-02; Study Completion 2005-10

PRIMARY OUTCOMES:
Rose Bengal staining

SECONDARY OUTCOMES:
Fluorescein staining
Total symptoms of dry eye
Tear break up time (TBUT)
Schirmer I test

CONTACTS AND LOCATIONS:
Overall Officials: Pitipong Suramethakul, MD, Study Director — Faculty of Medicine, Chulalongkorn University, Bangkok Thailand; Vilavun Puangsricharern, MD, Principal Investigator — Faculty of Medicine, Chulalongkorn University, Bangkok Thailand; Nipaporn Maneerat, MD, Study Director — Faculty of Medicine, Chulalongkorn University, Bangkok Thailand
Locations (1):
- Chulalongkorn Hospital, Bangkok, Bangkok, Thailand

REFERENCES:
- [Background] Schein OD, Munoz B, Tielsch JM, Bandeen-Roche K, West S. Prevalence of dry eye among the elderly. Am J Ophthalmol. 1997 Dec;124(6):723-8. doi: 10.1016/s0002-9394(14)71688-5. PMID 9402817
- [Background] Hikichi T, Yoshida A, Fukui Y, Hamano T, Ri M, Araki K, Horimoto K, Takamura E, Kitagawa K, Oyama M, et al. Prevalence of dry eye in Japanese eye centers. Graefes Arch Clin Exp Ophthalmol. 1995 Sep;233(9):555-8. doi: 10.1007/BF00404705. PMID 8543205
- [Background] Lee AJ, Lee J, Saw SM, Gazzard G, Koh D, Widjaja D, Tan DT. Prevalence and risk factors associated with dry eye symptoms: a population based study in Indonesia. Br J Ophthalmol. 2002 Dec;86(12):1347-51. doi: 10.1136/bjo.86.12.1347. PMID 12446361
- [Background] Brewitt H, Sistani F. Dry eye disease: the scale of the problem. Surv Ophthalmol. 2001 Mar;45 Suppl 2:S199-202. doi: 10.1016/s0039-6257(00)00202-2. PMID 11587143
- [Background] Bron AJ. Diagnosis of dry eye. Surv Ophthalmol. 2001 Mar;45 Suppl 2:S221-6. doi: 10.1016/s0039-6257(00)00201-0. PMID 11587146
- [Background] Sheppard JD. Guidelines for the treatment of chronic dry eye disease. Manag Care. 2003 Dec;12(12 Suppl):20-5. PMID 14723110
- [Background] Horwath-Winter J, Berghold A, Schmut O, Floegel I, Solhdju V, Bodner E, Schwantzer G, Haller-Schober EM. Evaluation of the clinical course of dry eye syndrome. Arch Ophthalmol. 2003 Oct;121(10):1364-8. doi: 10.1001/archopht.121.10.1364. PMID 14557170
- [Background] Noecker R. Effects of common ophthalmic preservatives on ocular health. Adv Ther. 2001 Sep-Oct;18(5):205-15. doi: 10.1007/BF02853166. PMID 11783457
- [Background] Albietz JM, Lenton LM, McLennan SG, Earl ML. A comparison of the effect of refresh plus and bion tears on dry eye symptoms and ocular surface health in myopic LASIK patients. CLAO J. 2002 Apr;28(2):96-100. PMID 12054380
- [Background] Noecker RJ. Comparison of initial treatment response to two enhanced-viscosity artificial tears. Eye Contact Lens. 2006 May;32(3):148-52. doi: 10.1097/01.icl.0000181819.63425.a6. PMID 16702870
- [Background] Sall K, Stevenson OD, Mundorf TK, Reis BL. Two multicenter, randomized studies of the efficacy and safety of cyclosporine ophthalmic emulsion in moderate to severe dry eye disease. CsA Phase 3 Study Group. Ophthalmology. 2000 Apr;107(4):631-9. doi: 10.1016/s0161-6420(99)00176-1. PMID 10768324
- [Background] Kojima T, Ishida R, Dogru M, Goto E, Matsumoto Y, Kaido M, Tsubota K. The effect of autologous serum eyedrops in the treatment of severe dry eye disease: a prospective randomized case-control study. Am J Ophthalmol. 2005 Feb;139(2):242-6. doi: 10.1016/j.ajo.2004.08.040. PMID 15733983
- [Background] S. Rozen, M. Ableson, A. Giovanoni, et al. Assessment of the comfort and tolerance of 0.5% carboxymethylcellulose preserved with purite (REFRESH TEARSTM) in dry eye sufferers. Invest Ophthalmol Vis Sci. 1998 Mar 15;39(4)S451.
- [Background] Peter J.McDonnell, John J.Doyle, Lee Stern, and The Dysfunctional Tear Syndrome Group